CLINICAL TRIAL: NCT00216957
Title: Randomized Clinical Trial Comparing Coronary Bypass Grafting With or Without Cardiopulmonary Bypass
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maritime Heart Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QE-RS/1998-220
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Coronary Artery Bypass; Cardiopulmonary Bypass

INTERVENTIONS:
Procedure: Coronary bypass surgery without cardiopulmonary bypass

SUMMARY:
Coronary artery bypass grafting (CABG) is a well established treatment modality for patients with coronary artery disease. For 30 years now CABG operations have been performed with the help of the heart lung machine (Cardiopulmonary bypass). However, the heart lung machine is believed to be responsible for many of the side effects and complications seen in patients following CABG surgery. The organs most commonly affected are the brain, blood constituents, lungs and kidneys.

In the last few years, stabilising devices have been developed that allow CABG operations to be performed safely without the use of the heart lung machine. Our hypothesis was that CABG done without the heart lung machine may be better tolerated by patients resulting in lower morbidity, increased functional outcome and shorter hospital length of stay.

Enrolment into the trial was from 1998 to 2003 and included 300 patients. The last patient was enrolled in June of 2003. The initial results from the study suggest that excellent results can be obtained with both techniques and contrary to others no advantages could be demonstrated in in-hospital outcomes of patients performed without cardiopulmonary bypass (Legare et al. Circulation 2005).

DETAILED DESCRIPTION:
We are now in follow-up to evaluate the medium term and long term outcomes of all 300 patients originally enrolled in above mentioned randomized clinical trial. The follow-up of patients is approved by the Capital Health Research Ethics Board (CDHA-RS/2004-295).

ELIGIBILITY:
Inclusion Criteria:

* Any patient suitable for CABG surgery

Exclusion Criteria:

* Emergency, concomitant procedure, low ejection fraction (<20%)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1998-10; Study Completion 2004-06

PRIMARY OUTCOMES:
Length of hospitalization
Blood product utilization
Post operative atrial fibrillation

SECONDARY OUTCOMES:
Myocardial infarction
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Legare, MD, Principal Investigator — Dalhousie University
Locations (1):
- Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia, Canada